CLINICAL TRIAL: NCT05510102
Title: Characterization of Medical Student Burnout Using Remote Physiologic Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Alexander Hajduczok, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21D.754
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Wellness; Burnout; Remote Monitoring
Keywords: WHOOP strap 4.0
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a treatment group (full remote monitoring data) versus a control arm (blinded data).
Who Masked: Investigator
Masking Description: Investigators are blinded to subject intervention group (data blinded versus data unblinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group (Experimental): Subjects will have full remote monitoring data access throughout the entirety of the study (6 months).
  Interventions: Device: WHOOP strap 4.0 (full data access)
- Control group (Active Comparator): Subjects will be blinded to remote monitoring data for the first 3 months of the study followed by an unblinding and full access to remote monitoring data at the 3 month mark (continued for the remainder of the study).
  Interventions: Device: WHOOP strap 4.0 (partial data access)

INTERVENTIONS:
Device: WHOOP strap 4.0 (full data access) — The WHOOP strap 4.0 provides continuous physiologic data via remote monitoring. Subjects will have full remote monitoring data access throughout the entirety of the study (6 months).
  Arms: Treatment group
Device: WHOOP strap 4.0 (partial data access) — The WHOOP strap 4.0 provides continuous physiologic data via remote monitoring. Subjects will be blinded to remote monitoring data for the first 3 months of the study followed by an unblinding and full access to remote monitoring data at the 3 month mark (continued for the remainder of the study).
  Arms: Control group

SUMMARY:
A reliable method for monitoring stress and burnout among medical students is critically needed. To address this gap, our team aims to utilize the cost-effective WHOOP strap 4.0 wearable device to continuously capture stress-relevant physiologic data (i.e., sleep hours, heart rate variability, respiration rate, resting heart rate) among up to 50 third-year medical students at 24 Sidney Kimmel Medical College at Thomas Jefferson University for 6 months.

DETAILED DESCRIPTION:
Aim 1: To determine whether physiologic metrics of sleep and heart rate variability correlate with subjective assessments of medical student wellness in a 6-month period.

Hypothesis: Less total sleep hours will correlate with higher scores for Perceived Stress Scale-4, Medical Student Well-Being Index, and Patient Health Questionnaire-9, but lower heart rate variability will correlate with higher scores on Perceived Stress Scale-4, Medical Student Well Being Index, and Patient Health Questionnaire-9.

Aim 2: To determine whether physiologic metrics of sleep and heart rate variability correlate with performance on shelf examinations for clinical rotations in a 6-month period.

Hypothesis: Less total sleep hours and lower heart rate variability will correlate with poorer performance on shelf examinations.

ELIGIBILITY:
Inclusion Criteria:

* Third-year medical student at Thomas Jefferson University
* ≥18 years of age
* Actively participating in family medicine, internal medicine, neurology, obstetrics/gynecology, pediatrics, psychiatry, surgery, or emergency medicine rotations
* Own a smart phone for Bluetooth pairing with WHOOP strap 4.0

Exclusion Criteria:

* Allergies, contraindications, or unwillingness to wear a wrist device for the study period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Total sleep hours per night | 180 days
  Sleep (hours per night) will be objectively measured nightly.
Medical Student Well-Being Index (MSWBI) | 180 days
  The MSWBI consists of 7 items, scored 0-7, with lower scores indicative of better medical student wellbeing. This survey will be administered biweekly.

SECONDARY OUTCOMES:
REM sleep hours, nightly | 180 days
  REM sleep hours will be measured nightly by the WHOOP strap 4.0.
Deep sleep hours, nightly | 180 days
  Deep sleep hours will be measured nightly by the WHOOP strap 4.0.
Resting heart rate, nightly | 180 days
  Resting heart rate will be measured nightly by the WHOOP strap 4.0.
Heart rate variability, nightly | 180 days
  Heart rate variability will be measured nightly by the WHOOP strap 4.0.
Respiration rate, nightly | 180 days
  Respiration rate will be measured nightly by the WHOOP strap 4.0.
Pulse oximetry, nightly | 180 days
  Pulse oximetry will be measured nightly by the WHOOP strap 4.0.
Body temperature, nightly | 180 days
  Body temperature will be measured nightly by the WHOOP strap 4.0.
Average duty hours per week | 180 days
  Duty hours will be self-reported every week
Perceived Stress Scale-4 | 180 days
  The PSS-4 consists of 4 items that assess perceived stress. The items are scored on a 4-point scale. This survey will be administered biweekly.
Patient Health Questionnaire-9 (PHQ-9) | 180 days
  The (Patient Health Questionnaire-9) PHQ-9 consists of 9 items that assess major depressive disorder. This survey will be administered biweekly. It is scored on a 0-27 scale with 27 representing most severe depression (worse outcomes).
Scores on shelf examinations | 180 days
  Subjects will self-report examination scores for shelf exams administered after each clinical rotation. Scores are reported on a 0-100 scale with 100 being the best score possible.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hajduczok, MD, Principal Investigator — Thomas Jefferson University Hospital, Department of Cardiology
Locations (1):
- Sidney Kimmel Medical College at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No